CLINICAL TRIAL: NCT03288714
Title: A Prospective, Multicenter, Double-Blind, Sham-Controlled Adaptive Design Study to Confirm the Safety and Efficacy of NEST sTMS in Subjects With Major Depressive Disorder Who Have Not Responded to at Least One Antidepressant Medication in the Current Episode
Brief Title: Adaptive Design Study of NEST sTMS in Subjects With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NND-3002
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major; Depressive Episode; Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation; TMS; sTMS
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Sham Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active sTMS (Experimental): Synchronized Transcranial Magnetic Stimulation (sTMS) treatments to be administered using an active device 5 times per week for six treatment weeks.
  Interventions: Device: Synchronized Transcranial Magnetic Stimulation (sTMS)
- Sham Stimulation (Sham Comparator): Sham treatments to be administered using a sham device 5 times per week for six treatment weeks.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Synchronized Transcranial Magnetic Stimulation (sTMS) — sTMS delivers brain stimulation via a continuous magnetic field created by the device and set to the individual patient's intrinsic alpha frequency (IAF).
  Arms: Active sTMS
Device: Sham Stimulation — Sham stimulation is designed to look, sound and feel like the investigational device, but does not deliver magnetic stimulation to the brain.
  Arms: Sham Stimulation

SUMMARY:
This is a double-blind, sham controlled, multi-center study to confirm the safety and efficacy of synchronized transcranial magnetic stimulation (sTMS) for the treatment of patients currently experiencing an episode of depression who have failed to respond to at least one (1) antidepressant medication. Patients will be randomly assigned to either active or sham therapy and will undergo daily treatments for a period of time. Following completion of blinded treatments, patients may be eligible for a course of open label treatments.

DETAILED DESCRIPTION:
Prospective, randomized, double-blind, sham-controlled, parallel group adaptive design study to confirm the safety and efficacy of sTMS in subject with Major Depressive Disorder (MDD) who have not responded to at least one antidepressant medication in the current episode. MDD was diagnosed according to DSM-IV criteria rendered by structured interview using the Mini International Neuropsychiatric Interview (MINI).

Subjects must have discontinued any antidepressant medication a minimum of 1 week prior to initiation of treatment with the active sTMS or sham device. Following wash-out of the antidepressant medication, an additional evaluation was performed to determine whether the protocol eligibility criteria were met before randomization and treatment.

Randomized subjects were treated 5 days per week for 6 weeks. Subjects who completed 6 weeks of double-blind treatment may have been eligible to receive up to 6 weeks of open-label treatment as clinically indicated during the follow-up phase of the study.

Follow-up evaluation visits were conducted during those six weeks, with frequency of the visits determined by the treatment choice during that time frame (open label subjects had weekly evaluation visits for 6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Current episode of Major Depressive Disorder
* Inadequate response to at least one antidepressant medication in the current episode (Treatment Resistant Depression)
* Investigator able to identify IAF using EEG
* Willingness and ability to adhere to treatment schedule (5 treatments per week for six weeks)

Exclusion Criteria:

* Unable to unwilling to give informed consent
* Diagnosed with excluded conditions or treatment histories
* Currently hospitalized due to severity of depression symptoms
* Use of prohibited medications (as defined by protocol) within specified time frame of randomization
* Use of certain cardiac devices
* Use of certain intracranial devices
* Currently pregnant or unwilling to practice acceptable means of birth control, and women who are breastfeeding

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Leuchter, MD, Principal Investigator — University of California, Los Angeles
Locations (14):
- United States (14):
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - UCLA Westwood - Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - New York University, New York, New York
  - Laureate Institute for Brain Research, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brain Health Consultants, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local referral networks, as well as online study descriptions, printed flyers, and radio advertisements approved by Institutional Review Boards (IRB). Recruitment was accomplished through initial interview and in-person screening assessments determining eligibility.
Pre-assignment Details: Following enrollment and completion of informed consent, participants were randomized to a treatment arm. Participants were instructed to discontinue any current antidepressant medication a minimum of 1 week prior to initiation of treatment, and confirmation of eligibility was completed after the wash-out.
Period: Overall Study
Arm/Group | Active sTMS | Sham Stimulation
Started | 59 | 62
Completed | 49 | 59
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Non-compliance with study schedule | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Clinical Worsening | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics taken from the per-protocol (PP) population; the PP group includes all participants who signed an informed consent, met study criteria, were randomized to a treatment arm, received at least 80% (24/30) of scheduled treatments within 60 days and completed the required treatment and post-baseline assessments in the double-blind phase
Groups:
- Total: Total of all reporting groups
Arm/Group | Active sTMS | Sham Stimulation | Total
Number analyzed (Participants) | 46 | 57 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.3) | 46.1 (13.0) | 45.6 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 43 | 75
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 6
  Black or African American | 4 | 4 | 8
  Hispanic | 4 | 5 | 9
  American Indian/Alaska Native | 0 | 1 | 1
  White | 34 | 44 | 78
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 57 | 103
Education Level [Count of Participants; unit: Participants]
  Some high school or less | 0 | 1 | 1
  High school diploma | 2 | 3 | 5
  Vocational school | 3 | 0 | 3
  Some college | 15 | 12 | 27
  College degree | 15 | 25 | 40
  Professional or graduate degree | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinical Response (Reduction of At Least 50% in Baseline HAMD-17 Score) in Per-Protocol Population
Description: Number of participants at the end of each treatment week who saw a reduction of at least 50% in baseline Hamilton Depression Rating Scale (HAMD-17) scores from baseline to week 6, compared between the active treatment and sham-controlled groups.
  The Hamilton Depression Rating Scale (HAMD-17) system asks 17 questions to rank subject on a scale ranges between 0-52, with higher numbers indicating more severe symptoms. 0-7 is generally accepted to be within the normal range (or in remission), while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Baseline (Day 0) to End of Weeks 1, 2, 3, 4, 5, 6
Population: 121 subjects were randomized into the study. Of those, 13 subjects dropped out of the study for various reasons and 5 were excluded from per-protocol analysis, as they failed to meet protocol requirements. Per-protocol analysis was performed on the remaining 103 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Active sTMS | Sham Stimulation
Number analyzed (Participants) | 46 | 57
Participants
  Week 1 | 5 | 2
  Week 2 | 7 | 10
  Week 3 | 9 | 12
  Week 4 | 11 | 10
  Week 5 | 12 | 16
  Week 6 | 11 | 12
Statistical Analysis 1: Comparison: Active sTMS vs Sham Stimulation; Null hypothesis is that the active sTMS treatment group does not differ from the sham group with respect to the proportion of patients with clinical response at Week 6; Test type: Superiority; p = .814, Fisher Exact; The proportion of patients is compared across treatment groups using Fisher's Exact

2. Secondary Outcome: Mean Change (SD) in HAMD-17 Scores From Baseline to End of Treatment
Description: Change from the baseline in HAMD-17 total score from baseline to week 6, compared between the active treatment and sham-controlled groups.
  The Hamilton Depression Rating Scale (HAMD-17) system asks 17 questions to rank subject on a scale ranges between 0-52, with higher numbers indicating more severe symptoms. 0-7 is generally accepted to be within the normal range (or in remission), while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Baseline (Day 0) and End of Weeks 1, 2, 3, 4, 5, 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on HAMD-17 scale
Arm/Group | Active sTMS | Sham Stimulation
Number analyzed (Participants) | 46 | 57
score on HAMD-17 scale
  Baseline | 22.96 (2.81) | 22.04 (4.01)
  Change from Baseline to Week 1 | -5.30 (5.14) | -4.33 (3.60)
  Change from Baseline to Week 2 | -6.63 (4.99) | -6.65 (4.93)
  Change from Baseline to Week 3 | -7.76 (5.48) | -7.74 (5.54)
  Change from Baseline to Week 4 | -7.61 (5.63) | -7.93 (6.19)
  Change from Baseline to Week 5 | -7.93 (5.81) | -7.95 (6.56)
  Change from Baseline to Week 6 | -7.57 (5.50) | -6.81 (6.48)
Statistical Analysis 1: Comparison: Active sTMS vs Sham Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .872, ANCOVA; P-value is from analysis of covariance adjusting for baseline

3. Secondary Outcome: Mean Change (SD) in MADRS Scores From Baseline to End of Treatment in the Per-Protocol Population
Description: Change from the baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score from baseline to week 6, compared between the active treatment and sham-controlled groups.
  The MADRS scale ranges between 0-54, with higher numbers indicating more severe symptoms. 0-6 is generally accepted to be within the normal range (or in remission), 7-19 represents mild depression, while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Baseline (Day 0) and End of Weeks 1, 2, 3, 4, 5, 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on MADRS scale
Arm/Group | Active sTMS | Sham Stimulation
Number analyzed (Participants) | 46 | 57
score on MADRS scale
  Baseline | 31.89 (4.57) | 30.72 (5.64)
  Change from Baseline to Week 1 | -6.02 (8.25) | -5.39 (5.80)
  Change from Baseline to Week 2 | -7.91 (7.46) | -8.63 (8.20)
  Change from Baseline to Week 3 | -10.76 (8.57) | -9.47 (9.19)
  Change from Baseline to Week 4 | -8.89 (9.81) | -10.12 (9.04)
  Change from Baseline to Week 5 | -9.11 (8.64) | -10.81 (8.88)
  Change from Baseline to Week 6 | -9.52 (8.75) | -9.77 (9.56)
Statistical Analysis 1: Comparison: Active sTMS vs Sham Stimulation; The null hypothesis is that the active sTMS treatment group does not differ; Test type: Superiority; p = .641, ANCOVA; P-value is from analysis of covariance adjusting for baseline

4. Secondary Outcome: Responder Analysis: Mean Change (SD) in HAMD-17 Scores From Baseline to End of Treatment in Per-Protocol Patients With Individual Alpha Frequency Greater Than 9.8 Hz
Description: Measure of change in mean (SD) of HAMD-17 scores from baseline to end of treatment in per-protocol patients with an Individual alpha frequency (IAF) of greater than 9.8Hz.
  The Hamilton Depression Rating Scale (HAMD-17) system asks 17 questions to rank subject on a scale ranges between 0-52, with higher numbers indicating more severe symptoms. 0-7 is generally accepted to be within the normal range (or in remission), while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Baseline (Day 0) and End of Weeks 1, 2, 3, 4, 5, 6
Population: Subjects in the per-protocol group with IAF greater than 9.8 Hz.
Measure: Mean (Standard Deviation); unit: score on HAMD-17 scale
Groups:
- Active sTMS (IAF > 9.8Hz): Synchronized Transcranial Magnetic Stimulation (sTMS) treatments to be administered using an active device 5 times per week for six treatment weeks.
  Synchronized Transcranial Magnetic Stimulation (sTMS): sTMS delivers brain stimulation via a continuous magnetic field created by the device and set to the individual patient's intrinsic alpha frequency (IAF), subgroup of those participants were found to be greater than 9.8Hz
- Sham Stimulation (IAF>9.8Hz): Sham treatments to be administered using a sham device 5 times per week for six treatment weeks.
  Sham Stimulation: Sham stimulation is designed to look, sound and feel like the investigational device, but does not deliver magnetic stimulation to the brain. All patients analyzed and compared with other belonging to same subgroup of those with IAF greater than 9.8Hz.
Arm/Group | Active sTMS (IAF > 9.8Hz) | Sham Stimulation (IAF>9.8Hz)
Number analyzed (Participants) | 19 | 33
score on HAMD-17 scale
  Baseline | 23.68 (2.65) | 21.91 (3.50)
  Change from Baseline to Week 1 | -7.05 (6.11) | -4.12 (3.32)
  Change from Baseline to Week 2 | -8.32 (5.75) | -6.15 (4.27)
  Change from Baseline to Week 3 | -10.11 (5.37) | -7.70 (4.22)
  Change from Baseline to Week 4 | -9.89 (4.74) | -6.97 (4.88)
  Change from Baseline to Week 5 | -9.53 (6.01) | -6.97 (6.14)
  Change from Baseline to Week 6 | -9.47 (5.11) | -5.18 (5.72)
Statistical Analysis 1: Comparison: Active sTMS (IAF > 9.8Hz) vs Sham Stimulation (IAF>9.8Hz); Test type: Superiority; p = .032, ANCOVA — Alpha level: .05; P-value is from analysis of covariance adjusting for baseline

5. Secondary Outcome: Mean Change (SD) in HAMD-17 Scores From Baseline to Week 6 of Open-Label Treatments
Description: Change in HAMD-17 total score during 6 weeks of open-label treatment, compared between the active treatment and sham-controlled groups.
  The Hamilton Depression Rating Scale (HAMD-17) system asks 17 questions to rank subject on a scale ranges between 0-52, with higher numbers indicating more severe symptoms. 0-7 is generally accepted to be within the normal range (or in remission), while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Baseline (sTMS Week 6/Sham Baseline) and End of Weeks 7, 8, 9, 10, 11, 12
Population: Of the 103 subjects in the original per-protocol group, 83 continued to open-label treatment for analysis.
Measure: Mean (Standard Deviation); unit: score on HAMD-17 scale
Arm/Group | Active sTMS | Sham Stimulation
Number analyzed (Participants) | 38 | 45
score on HAMD-17 scale
  sTMS Active Treatment Week 6/Sham Baseline | 16.50 (4.69) | 16.76 (5.35)
  Change from Baseline to Open-Label Week 1 (Active Week 7/Sham Week 1) | -8.82 (5.34) | -3.98 (5.53)
  Change from Baseline to Open-Label Week 2 (Active Week 8/Sham Week 2) | -9.36 (5.96) | -3.69 (5.17)
  Change from Baseline to Open-Label Week 3 (Active Week 9/Sham Week 3) | -9.09 (6.58) | -4.29 (5.25)
  Change from Baseline to Open-Label Week 4 (Active Week 10/Sham Week 4) | -10.68 (7.34) | -4.51 (5.92)
  Change from Baseline to Open-Label Week 5 (Active Week 11/Sham Week 5) | -12.34 (6.54) | -5.47 (5.71)
  Change from Baseline to Open-Label Week 6 (Active Week 12/Sham Week 6) | -12.72 (6.97) | -6.42 (5.01)
Statistical Analysis 1: Comparison: Active sTMS vs Sham Stimulation; Test type: Superiority; p = .015, ANCOVA — Alpha level: .05; P-value is from analysis of covariance adjusting for baseline

6. Secondary Outcome: Incidence of Clinical Response (Reduction of At Least 50% in Baseline HAMD-17 Score) in Open-Label Per-Protocol Population
Description: Number of participants seeing reduction of at least 50% in baseline Hamilton Depression Rating Scale (HAMD-17) scores during 6 weeks of open-label treatment, compared between the active treatment and sham-controlled groups.
  The Hamilton Depression Rating Scale (HAMD-17) system asks 17 questions to rank subject on a scale ranges between 0-52, with higher numbers indicating more severe symptoms. 0-7 is generally accepted to be within the normal range (or in remission), while a score of 20 or higher indicates moderate to severe depression.
Time Frame: Baseline (sTMS Week 6/Sham Baseline) and End of Weeks 7, 8, 9, 10, 11, 12
Population: Of the 103 subjects in the original per-protocol group, 83 continued to open-label treatment for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Active sTMS | Sham Stimulation
Number analyzed (Participants) | 38 | 45
Participants
  Open Label Week 1 (Active Week 7/Sham Week 1) | 12 | 9
  Open Label Week 2 (Active Week 8/Sham Week 2) | 17 | 9
  Open Label Week 3 (Active Week 9/Sham Week 3) | 14 | 10
  Open Label Week 4 (Active Week 10/Sham Week 4) | 19 | 10
  Open Label Week 5 (Active Week 11/Sham Week 5) | 23 | 10
  Open Label Week 6 (Active Week 12/Sham Week 6) | 20 | 12
Statistical Analysis 1: Comparison: Active sTMS vs Sham Stimulation; Test type: Superiority; p = .028, Fisher Exact — Alpha level: .05; The proportion of patients is compared across treatment groups using Fisher's Exact

ADVERSE EVENTS:
Time Frame: All subjects screened at Screening, Baseline, and each Evaluation Visit (End of Weeks 1, 2, 3, 4, 5, 6; if continuing open-label 7, 8, 9, 10, 11, 12)
Description: All adverse events were entered by study personnel verbatim based on patient reports.
  Any adverse event occurring before randomization occurred was not included in the final report.
Arm/Group | Active sTMS | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/59 | 0/62
Other Adverse Events (participants affected / at risk) | 35/59 | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active sTMS (N=59) | Sham Stimulation (N=62)
Hospitalization (Suicidal Ideation) (Psychiatric disorders) | 1 | 0 — Patient exhibited increased depressive symptoms and suicidal ideation and was subsequently admitted to the hospital for suicidal ideation.
Anaphylactic Reaction (peanut allergy) (General disorders) | 1 | 0 — Subject in Open-label portion of study had anaphylactic reaction to peanuts and was admitted to hospital for treatment. Subject continued treatment normally.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active sTMS (N=59) | Sham Stimulation (N=62)
Application Site Discomfort (Skin and subcutaneous tissue disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dizziness (General disorders) | 3 | 1
Headache (Nervous system disorders) | 23 | 28
Insomnia (Psychiatric disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 6 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Visual Disturbance (Eye disorders) | 3 | 5
Paraesthesia (Nervous system disorders) | 1 | 5
Anxiety (Psychiatric disorders) | 1 | 2
Cramping (General disorders) | 0 | 2
GI Infection (Gastrointestinal disorders) | 0 | 2
Oral Herpes (General disorders) | 2 | 0
Blepharospasm (General disorders) | 2 | 1
Hypersensitivity (General disorders) | 0 | 2
Jaw Discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Twitching (General disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Nasopharyngitis (General disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
* Sham device used exaggerated vibration at the IAF which may have provided active treatment in the form of trigeminal nerve stimulation
* Short wash-out period may have negatively impacted results.
* Short treatment duration may limit efficacy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT03288714/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT03288714/SAP_001.pdf